CLINICAL TRIAL: NCT01494714
Title: A Study to Evaluate Skin Irritation and Photo Irritation of JNJ 10229570-AAA on Intact Skin of Japanese Healthy Male Subjects
Brief Title: A Study to Evaluate Skin Irritation and Photo Irritation of JNJ 10229570-AAA on Intact Skin of Japanese Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: CR018670; 10229570-JPN-01 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2011-12-13; First posted 2011-12-19 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers; JNJ 10229570-AAA; Skin irritation; Skin photo irritation
MeSH Terms: interventions — Petrolatum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Closed-patch test (Experimental)
  Interventions: Drug: JNJ 10229570-AAA 1.2% cream; Drug: JNJ 10229570-AAA 2.4% cream; Drug: JNJ 10229570-AAA 3.6% cream; Drug: Color-matched vehicle in a cream formulation containing 0 mg of JNJ 10229570-AAA; Drug: Petroleum jelly

INTERVENTIONS:
Drug: JNJ 10229570-AAA 1.2% cream — A patch containing the cream will be applied on the back and left for 48 hours on the left side, and 24 hours on the right side.
Drug: JNJ 10229570-AAA 2.4% cream — A patch containing the cream will be applied on the back and left for 48 hours on the left side, and 24 hours on the right side.
Drug: JNJ 10229570-AAA 3.6% cream — A patch containing the cream will be applied on the back and left for 48 hours on the left side, and 24 hours on the right side.
Drug: Color-matched vehicle in a cream formulation containing 0 mg of JNJ 10229570-AAA — A patch containing the cream will be applied on the back and left for 48 hours on the left side, and 24 hours on the right side.
Drug: Petroleum jelly — A patch containing the petroleum jelly will be applied on the back and left for 48 hours on the left side, and 24 hours on the right side.

SUMMARY:
The purpose of this study is to evaluate skin irritation and photo irritation of JNJ 10229570-AAA on intact skin of Japanese healthy male participants.

DETAILED DESCRIPTION:
This is a single center, interpreter-blinded (the person interpreting the results does not know the name of the assigned drug), randomized (drug is assigned by chance like flipping a coin), vehicle-controlled, closed-patch test study. Thirty (30) Japanese participants will be enrolled in the study. Each treatment (JNJ 10229570-AAA at 1.2%, 2.4%, 3.6%, vehicle in a cream formulation, and petroleum jelly) will be randomly applied in vertical position on the back of each participant, with a corresponding strength applied at the same vertical position (left vs. right). The study drugs applied on the left side will be washed off at 48 hours after application. The dermatological evaluation and photo shoots will be done at 1 (T49) and 24 (T72) hours after washing off the drugs. All participants who completed the dermatological evaluation will be included in the evaluation of skin irritation and skin photo irritation. The study drugs applied on the right side will be washed off at 24 hours after application. The dermatological evaluation and photo shoots will be done at 1 hour after washing off. Ultraviolet A (UVA) will be irradiated to the application site. One hour after irradiation start (T26), the dermatological evaluation and photo shoots will be done. Afterwards the application site will be covered for the protection against UV. Twenty-four hours after washing off (T48), the cover will be taken off, and then the dermatological evaluation and photo shoots will be done at 1 (T49) and 24 (T72) hours. Additionally, the safety profile of JNJ 10229570-AAA will be assessed during the study. The study has a total duration of maximum 32 days.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent document
* Body mass index between 18.0 and 30.0 kg/m2 (inclusive), and body weight not less than 50 kg
* Blood pressure between 90 and 140 mmHg systolic (inclusive), and no higher than 90 mmHg diastolic
* Electrocardiogram (ECG) consistent with normal cardiac conduction and function
* Non-smoker
* Agree to use an adequate contraception method

Exclusion Criteria:

* History of or current clinically significant medical illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, biochemistry or urinalysis
* Clinically significant abnormal physical examination, vital signs or ECG
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements) within 14 days before the study treatment
* History of drug or alcohol abuse within the past 5 years
* Drug allergy or drug hypersensitivity
* Blood donation, depending on the volume of blood collection
* Positive test for human immunodeficiency virus (HIV), hepatitis B or C, or syphilis
* Dermatological disease at application site
* Photosensitivity
* Exposure to excessive or chronic ultraviolet (UV) radiation (i.e., sunbathing, tanning salon use, phototherapy) within 4 weeks prior to study treatment or planned during the study period

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Skin irritation according to the Japanese evaluation criteria (scores on a scale) | 72 hours
  The Japanese skin irritation evaluation criteria is a 6-point scale specifying the irritation level of the skin, from 0 (no response) to 4 (blister)
Skin photo irritation according to the Japanese evaluation criteria (scores on a scale) | 72 hours
  The Japanese skin photo irritation evaluation criteria is a 6-point scale specifying the level of skin photo irritation from 0 (lack of reaction or reaction comparable to non-irradiated site) to 4 (reaction four ranks more pronouced using domestic criteria compared with non-irradiated site)

SECONDARY OUTCOMES:
Skin irritation according to the International Contact Dermatitis Research Group (ICDRG) criteria (measurements on a scale) | 72 hours
  The ICDRG scale measures the level of skin irritation from Negative (no reaction) to Extreme Positive Reaction (erythema, infiltration, confluent vesicles)
Skin photo irritation according to the International Contact Dermatitis Research Group (ICDRG) criteria (measurements on a scale) | 72 hours
  The ICDRG scale measures the level of skin irritation from Negative (no reaction) to Extreme Positive Reaction (erythema, infiltration, confluent vesicles)
Number of participants with adverse events as a measure of safety and tolerability | 32 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (2):
- Japan (2):
  - Fukukoka
  - Hakata